CLINICAL TRIAL: NCT05553990
Title: Predictive Value of Human Microbiome and Serological Markers for Clinical Outcome of Acute Ischemic Stroke With Active Cancer
Brief Title: Predictive Value of Human Microbiome and Serological Markers for Clinical Outcome of AIS With Active Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2022-169
Record Dates: First submitted 2022-09-13; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Stroke, Acute; Tumor Progression
MeSH Terms: conditions — Ischemic Stroke; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, oral swabs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute ischemic stroke with active tumor: Acute ischemic stroke with active tumor
  Interventions: Other: intestinal flora disturbance
- Acute ischemic stroke without active tumor: Acute ischemic stroke without active tumor

INTERVENTIONS:
Other: intestinal flora disturbance — To observe the clinical prognosis of stroke patients complicated with tumor after enterobacterial disorder
  Groups: Acute ischemic stroke with active tumor

SUMMARY:
Explore with active cancer patients with acute ischemic stroke in the human body characteristic microorganism disorder to clinical prognosis of the predictive value of the secondary objective: to observe with active cancer patients with acute ischemic stroke in the body of microorganisms and their serological indexes change law of exploration condition change related biomarkers of microscopic objects group based on the human body.

DETAILED DESCRIPTION:
investigators recently found that changes in gut microbiota in patients with ischemic stroke are associated with the development of disease. However, there are few studies on the correlation between ischemic stroke with cancer and human microbiome and metabolites Whether the human microbiome and its metabolites are associated with the prognosis of such patients remains to be investigated. Therefore, this study hypothesized that structural changes in the human microbiome and its metabolites in patients with acute ischemic stroke with active cancer were associated with stroke severity and disease recovery Therefore, this topic proposed by collecting active follow-up cancer of acute ischemic stroke patients after admission and oral swabs Excrement and urine and blood samples, and based on the queue, follow-up analysis of the human microbiome dynamic change rule and the prognosis of patients with cancer of the acute ischemic stroke correlation, activity, further explore the secondary prevention of stroke management strategy based on the human microbiome.

ELIGIBILITY:
Inclusion Criteria:

* 1: It meets the diagnostic criteria for acute ischemic stroke

  2: Age ≥ 18 years

  3: The onset time is less than or equal to 2 weeks

  4: Diagnosis of cancer before stroke onset or during hospitalization and active cancer (failure to meet clinical criteria for cure, or discovery of recurrence or metastasis)

  5: Sign an informed consent form, provide relevant medical history information and provide biological specimens

Exclusion Criteria:

* 1: Previous history of disabling stroke (pre-onset mRS ≥2)

  2: Primary central nervous system tumor or hematologic system tumor

  3: The cancer meets the criteria for clinical cure and has not recurred or metastasized for more than 5 years

  4: Antibiotics, prebiotics/probiotics taken within 1 month

  5: Patients who cannot have stool specimens within 4 days of admission

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke with active tumor
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-06-07 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Neurological function score (mRS score) | 3 months after onset
  Neurological function score (mRS score) ，The minimum score is 0 and the maximum score is 5，The higher the mRS score, the worse the prognosis
Mortality | 3 months after onset
  Mortality

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale score(NIHSS score) | The first and seventh days of hospitalization、3 months, 6 months and 12 months after onset
  National Institutes of Health Stroke Scale score(NIHSS score) ，The minimum score is 0 and the maximum score is 42，The higher the NIHSS score, the worse the neurological function
Barthel Index | 3 months, 6 months and 12 months after onset
  Barthel Index，The minimum score is 0 and the maximum score is 100，The higher the BI index, the better the ability to take care of yourself
Mini-mental State Examination | Seventh day of hospitalization、3 months and 6 months after onset
  Mini-mental State Examination，The minimum score is 0 and the maximum score is 30，Closely related to educational attainment, the higher the score, the better the Closely related to educational attainment, the higher the score, the better the Closely related to educational attainment, the higher the score, the better the cognitive function
Montreal Cognitive Assessment | Seventh day of hospitalization、3 months and 6 months after onset
  Montreal Cognitive Assessment，The minimum score is 0 and the maximum score is 30，Closely related to educational attainment, the higher the score, the better the cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: JIA YIN, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong, China